CLINICAL TRIAL: NCT02979990
Title: Learning From Online Video Education for Controlled Ovarian Stimulation
Acronym: LOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-20821
Record Dates: First submitted 2016-11-09; First posted 2016-12-02 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Self Efficacy
Keywords: infertility; education
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Video (Placebo Comparator): Subjects will have access to general videos on the in vitro fertilization process. They will not have access to instructional videos related to the administration of controlled ovarian stimulation.
  Interventions: Other: Control Video
- Experimental Video (Experimental): Subjects will be asked to view instructional videos related to the administration of controlled ovarian stimulation medication during their own controlled ovarian stimulation
  Interventions: Other: Instructional Video

INTERVENTIONS:
Other: Instructional Video — The experimental group will be asked to view a set of videos that demonstrate proper usage of controlled ovarian stimulation medication. They will have the opportunity to review instructional videos as needed throughout the ovarian stimulation process.
  Arms: Experimental Video
Other: Control Video — The control group will have access to a video about the IVF process
  Arms: Control Video

SUMMARY:
The Learning from Online Video Education (LOVE) study seeks to determine if online instructional videos on how to administer medication needed for in vitro fertilization (IVF) help improve the quality of life and reduce stress during the IVF process.

DETAILED DESCRIPTION:
The Learning from Online Video Education (LOVE) is a randomized controlled trial that seeks to determine the effect of instructional online videos on medication administration on psychological well being during controlled ovarian stimulation.

The investigators hypothesize that usage of online instructional videos by women undergoing their first cycle of controlled ovarian stimulation for in vitro fertilization or oocyte cryopreservation improves measures of psychological well-being (Infertility Self Efficacy Scale, FertiQoL-T and Perceived stress scores) when compared to subjects that do not have access to this educational resource.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing first controlled ovarian stimulation cycle at the time of enrollment
* Has internet access

Exclusion Criteria:

* Had prior controlled ovarian stimulation cycle
* Does not have internet access
* Declines in person IVF medication teaching session
* Treating physician requests that patient not be approached for participation (any reason)

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 368 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Infertility Self Efficacy Scale | The infertility self efficacy scale score will be collected up to two weeks after egg retrieval
  Short questionnaire to determine a subjects self efficacy related to fertility treatment

SECONDARY OUTCOMES:
FertiQoL-T score | The Ferti-QoL-T score will be collected up to two weeks after egg retrieval
  The FertiQoL-T questionnaire is a previously validated instrument to assess ones quality of life as it relates to the administration of fertility medication administration.
Perceived stress score | The perceived stress score will be collected up to two weeks after egg retrieval
  This is a well validated psychological instrument used to measure one's perception of stress

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gameiro S, Boivin J, Peronace L, Verhaak CM. Why do patients discontinue fertility treatment? A systematic review of reasons and predictors of discontinuation in fertility treatment. Hum Reprod Update. 2012 Nov-Dec;18(6):652-69. doi: 10.1093/humupd/dms031. Epub 2012 Aug 6. PMID 22869759
- [Background] Omurtag K, Jimenez PT, Ratts V, Odem R, Cooper AR. The ART of social networking: how SART member clinics are connecting with patients online. Fertil Steril. 2012 Jan;97(1):88-94. doi: 10.1016/j.fertnstert.2011.10.001. Epub 2011 Nov 14. PMID 22088209
- [Background] Cousineau TM, Lord SE, Seibring AR, Corsini EA, Viders JC, Lakhani SR. A multimedia psychosocial support program for couples receiving infertility treatment: a feasibility study. Fertil Steril. 2004 Mar;81(3):532-8. doi: 10.1016/j.fertnstert.2003.08.021. PMID 15037398
- [Background] Turner K, Reynolds-May MF, Zitek EM, Tisdale RL, Carlisle AB, Westphal LM. Stress and anxiety scores in first and repeat IVF cycles: a pilot study. PLoS One. 2013 May 23;8(5):e63743. doi: 10.1371/journal.pone.0063743. Print 2013. PMID 23717472
- [Background] Garcia D, Vassena R, Prat A, Vernaeve V. Increasing fertility knowledge and awareness by tailored education: a randomized controlled trial. Reprod Biomed Online. 2016 Jan;32(1):113-20. doi: 10.1016/j.rbmo.2015.10.008. Epub 2015 Oct 30. PMID 26611499
- [Derived] Adeleye A, Cruz K, Cedars MI, Pasch L, Huddleston H. Learning from Online Video Education (LOVE) improves confidence in fertility treatments: a randomized controlled trial. NPJ Digit Med. 2022 Aug 29;5(1):128. doi: 10.1038/s41746-022-00673-y. PMID 36038614
- [Derived] Adeleye A, Cruz K, Pasch L, Huddleston H. Differences in perceived stress during ovarian stimulation between women with infertility and those pursing oocyte cryopreservation. Fertil Steril. 2020 Nov;114(5):1076-1084. doi: 10.1016/j.fertnstert.2020.05.025. Epub 2020 Aug 18. PMID 32826049